CLINICAL TRIAL: NCT03818373
Title: Can Ventilatory Response at Rest Predict Ventilatory Efficacy and Exercise Tolerance in Patients With a Univentricular Congenital Heart Disease?
Brief Title: Respiratory Drive in Patients With Univentricular Congenital Heart Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RECHMPL17_0400; UF 7512 (Other: Montpellier University hospital)
Record Dates: First submitted 2019-01-24; First posted 2019-01-28 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2021-12

CONDITIONS: Univentricular Heart; Children, Adult
Keywords: Univentricular congenital heart; Sleep apnea; Polysomnography; Respiratory drive; VE/VCO2 slope
MeSH Terms: conditions — Univentricular Heart; Sleep Apnea Syndromes

STUDY DESIGN:
Intervention Model Description: all participants receive the same intervention throughout the protocol
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with univentricular congenital heart disease (Other): Patients 8 years old or more with functionally univentricular congenital heart disease
  Interventions: Procedure: polysomnography

INTERVENTIONS:
Procedure: polysomnography — Sleep examination strictly non-invasive with skin sensors. This exploration would allow for the detection of respiratory sleep disorders and consider of appropriate management for patients.

SUMMARY:
The aim is to evaluate the correlation between the respiratory control to hypercapnia at rest and the VE/VCO2 slope measured during cardiopulmonary exercise testing.

The hypothesis is that patient with univentricular congenital heart disease have a increasing of respiratory drive like chronic heart failure. This increasing of respiratory drive could participate in the increasing of VE/VCO2 slope measured during cardiopulmonary exercise testing and in the genese of central apnea index during the sleep.

DETAILED DESCRIPTION:
The patients with univentricular congenital heart disease will perform :

* a cardiopulmonary exercise testing with measure VE/VCO2 slope,
* a measure of the respiratory drive to hypercapnia with occlusion pressure during the rebreathing with at rest (P0,1/PetCO2).
* A polysomnography with a scoring of central apnea index. Correlation will be evaluate between P 0,1/PetCO2 with VE/VCO2 slope and between P0,1/PetCO2 central apnea index.

ELIGIBILITY:
Inclusion Criteria:

* Functionally univentricular congenital heart disease
* Age ≥ 8 years
* Consent of the adult patient or the parents or legal guardians of the minor patient.
* Beneficiary of the social security scheme

Exclusion Criteria:

* Size <120 cm (minimum size for the stress test)
* Medical contraindication to exercise test or presence of : myocardial infarction less than 3 months old, unstable angina, uncontrolled severe arrhythmias, symptomatic aortic stenosis, uncontrolled heart failure, pulmonary embolism, evolutionary phlebitis, pericarditis, myocarditis, progressive endocarditis, aortic dissection
* Unstable patient with severe intellectual disability or complex pathology making polysomnography impossible
* Pregnant woman

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2021-07-07 (Actual); Study Completion 2021-07-07 (Actual)

PRIMARY OUTCOMES:
Pearson correlation - The measure the respiratory drive to hypercapnia with P0.1 during the rebreathing technique at rest | day 90 after inclusion visit (visit 2)
  between the measure the respiratory drive to hypercapnia with P0.1 during the rebreathing technique at rest
  - between VE/VCO2 slope during a cardiopulmonary exercise

SECONDARY OUTCOMES:
Pearson correlation | day 90 after inclusion visit (visit 2)
  * between the measure of the respiratory drive to hypercapnia with P0.1, the rebreathing technique at rest and Central apnea index scored with a polysomnography during a night
  * between the measure of the respiratory drive to hypercapnia with P0.1, the rebreathing technique at rest and NYHA, New York Heart Association Functional Classification
  * between the measure of the respiratory drive to hypercapnia with P0.1, the rebreathing technique at rest and the quality of life evaluated by questionary
  * between the measure of the respiratory drive to hypercapnia with P0.1, the rebreathing technique at rest and data of cardiac echography

CONTACTS AND LOCATIONS:
Overall Officials: Johan MOREAU, Principal Investigator — Montpellier University Hospital
Locations (2):
- France (2):
  - Arnaud de Villeneuve - University Hospital Pediatric and Congenital Cardiology Department Regional Reference Center - M3C, Montpellier, Occitanie
  - Institut Saint-Pierre, Palavas-les-Flots